CLINICAL TRIAL: NCT03545529
Title: Medico-economic Assessment of a "IsereADOM" Package of Services Versus Conventional Monitoring in the Care of a Population of Frail Elderly People With Loss of Autonomy.
Brief Title: Clinical and Medico-economic Evaluation of the Cohort "People at Risk of Falling"
Acronym: PARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC16.044
Record Dates: First submitted 2018-02-28; First posted 2018-06-04 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Fall Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Innovative supported (Experimental): In addition to usual care, patients benefit from connected tools (telealarm, numeric communication diary...) and from a strong accompaniment with a referent person who help better the patient.
  Interventions: Other: Innovativ supported
- conventional supported (No Intervention): Patients benefit from usual care

INTERVENTIONS:
Other: Innovativ supported — addition of connected tools and stronger accompaniment to prevent falls
  Arms: Innovative supported

SUMMARY:
The goal of this study is to evaluate the effectiveness of the IsereADOM service package compared to conventional follow-up on the risk of recurrence of falls at 6 months in frail elderly subjects.

There is a medico-economic goal too, is to conduct a cost-utility analysis of the IsereADOM service bundle compared to conventional 6-month follow-up from the community perspective in the cheat population at risk of re-offending.

ELIGIBILITY:
Inclusion Criteria :

* Patient falling at least 2 times in the year preceding the inclusion, one of them has been reported or consulted by a health care service ;
* Patient fragile and loss of autonomy: level of dependence with GIR 3, 4 and 5 ;
* Patient domiciled in the department of Isère ;
* Patient who can be followed regularly for 6 months ;
* Patient benefiting from an assistance plan : APA, PAP, CARSAT ;
* Patient affiliated with social security or beneficiary of such a scheme ;
* Patient able to read, write and understand French ;
* Patient having signed informed consent to participate.

Exclusion Criteria :

* Patient without professional or family carer of proximity ;
* Patient with moderate to severe cognitive impairment defined by MMS <23 ;
* Patient residing in a nursing home or institution for dependent person ;
* Persons referred to in Articles L1121-5 to L1121-8 of the CSP (corresponds to all persons protected: pregnant woman, parturient, mother who is breastfeeding, person deprived of liberty by judicial or administrative decision, person subject of a legal protection measure).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-10-12 (Actual)

PRIMARY OUTCOMES:
comparison of the number of falls according to the innovative or non-innovative care of frail elderly people | 6 months
  The outcome measure is the number of falls with hospitalization collected through administrative data from health facilities

CONTACTS AND LOCATIONS:
Overall Officials: Pascal COUTURIER, MD, Principal Investigator — CHU Grenoble Alpes
Locations (3):
- France (3):
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - CHU Grenoble-Alpes, Grenoble
  - Centre Hospitalier de Voiron, Voiron

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Sherrington C, Gates S, Clemson LM, Lamb SE. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2012 Sep 12;2012(9):CD007146. doi: 10.1002/14651858.CD007146.pub3. PMID 22972103
- [Background] Moyer VA; U.S. Preventive Services Task Force. Prevention of falls in community-dwelling older adults: U.S. Preventive Services Task Force recommendation statement. Ann Intern Med. 2012 Aug 7;157(3):197-204. doi: 10.7326/0003-4819-157-3-201208070-00462. PMID 22868837
- [Background] Gates S, Smith LA, Fisher JD, Lamb SE. Systematic review of accuracy of screening instruments for predicting fall risk among independently living older adults. J Rehabil Res Dev. 2008;45(8):1105-16. PMID 19235113
- [Background] Payen JF, Chanques G, Mantz J, Hercule C, Auriant I, Leguillou JL, Binhas M, Genty C, Rolland C, Bosson JL. Current practices in sedation and analgesia for mechanically ventilated critically ill patients: a prospective multicenter patient-based study. Anesthesiology. 2007 Apr;106(4):687-95; quiz 891-2. doi: 10.1097/01.anes.0000264747.09017.da. PMID 17413906
- [Background] Manca A, Hawkins N, Sculpher MJ. Estimating mean QALYs in trial-based cost-effectiveness analysis: the importance of controlling for baseline utility. Health Econ. 2005 May;14(5):487-96. doi: 10.1002/hec.944. PMID 15497198
- See also: Repérage et maintien de l'autonomie des personnes agées fragiles — http://www.fragilite.org